CLINICAL TRIAL: NCT04009785
Title: Evaluation of the Prevalence of Anti-infective Drug Compliance in Pediatric Patients Hospitalized at Nimes University Hospital After Return Home
Acronym: PEDIAOBST
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Mobilité/2017/GLB; 2017-A03114-49 (Other: ANSM)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Anti Infective; Pediatric Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, resistance to anti-infectives has become a global public health problem and its increased prevalence threatens human health.

To date, few studies have focused on drug compliance in the paediatric population and it varies according to the pathology This drug adherence in the paediatric population is directly linked to outpatient care by the parents or the child's immediate family. In addition, there are no studies on adherence to antibiotics prescribed at the end of hospitalization in the paediatric population.

In this context, it seems urgent to seek an intervention capable of leading to responsible and appropriate use of antibiotics in order to improve efficiency in the drug management of acute paediatric infections.

This pilot study would characterize pediatric patients and determine the compliance rate in this population.

ELIGIBILITY:
Inclusion Criteria:

* The patient is under 16 years of age (< 16 years of age).
* The patient is admitted to a full hospitalization in one of the 2 paediatric units of the University Hospital of Nîmes.
* The patient is discharged with a prescription for anti-infectives to be taken at home, for a maximum of 30 days.
* The patient and the holder of parental authority are available for a follow-up of 1 month after discharge from hospital.

Exclusion Criteria:

-

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients included in the study are patients under 16 years of age (< 16 years of age) admitted to full hospitalization in the paediatric units
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Rate of patients observing anti-infectives | 2018

SECONDARY OUTCOMES:
Rehospitalization rates / emergency visits related to worsening infection | 2018

OTHER OUTCOMES:
Rate of observing patients who have recovered their anti-infective treatment | 2018
Rate of observing patients who have taken anti-infective treatment as prescribed | 2018
Sociodemographic and clinical characteristics | 2018
Overall success rate in the quiz on understanding anti-infectives | 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nimes, Nîmes, France

REFERENCES:
- [Result] Warembourg M, Lonca N, Filleron A, Tran TA, Knight M, Janes A, Soulairol I, Leguelinel-Blache G. Assessment of anti-infective medication adherence in pediatric outpatients. Eur J Pediatr. 2020 Sep;179(9):1343-1351. doi: 10.1007/s00431-020-03605-8. Epub 2020 Mar 5. PMID 32140853